CLINICAL TRIAL: NCT05282667
Title: Significance of Barrier Membrane in the Reconstructive Management of Peri-implantitis: A RCT
Brief Title: Reconstructive Management of Peri-implantitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center of Implantology, Oral and Maxillofacial Surgery, Badajoz, Spain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2021-09-12; First posted 2022-03-16 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Resolution of Pathologic Process

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resorbable cross-linked barrier membrane (Experimental): Bone graft will be covered with a resorbable barrier membrane to exclude undesired cells from the area aimed at being regenerated (peri-implantitis bone defect)
  Interventions: Procedure: Reconstructive therapy of peri-implantitis by means of bone graft (and barrier membrane in the test group)
- No barrier membrane (Experimental): Bone graft will be solely packed in the peri-implantitis bone defect with no membrane to cover
  Interventions: Procedure: Reconstructive therapy of peri-implantitis by means of bone graft (and barrier membrane in the test group)

INTERVENTIONS:
Procedure: Reconstructive therapy of peri-implantitis by means of bone graft (and barrier membrane in the test group) — A full-thickness flap was raised to ensure sufficient access. Debridement of granulation tissue was subsequently conducted using a "mini-five" curette (Hu-Friedy) and site-specific Gracey curettes (Hu-Friedy). The surgical approach was tailored to the clinical scenario. Specifically, resective therapy by means of implantoplasty was performed for supracrestal defects (Meisinger LLC, Nauss, Germany). Surface detoxification was performed with 3% hydrogen peroxide during 2 minutes and irrigation with 0.12% chlorhexidine. The intraosseous compartment was grafted using mineralized and demineralized bone graft (LifeNet Health, Virginia, USA). The graft was compartmentalized in the test group with a collagen porcine resorbable membrane (RTM, Cytoplast, California, USA) adapted to the defect morphology. Nylon 5.0 (Resorba Sutures, Osteogenics Biomedical, Lubbock, Texas) was used for suturing, ensuring primary wound closure

SUMMARY:
With the growing burden of peri-implantitis around the globe, interest has flourished on the management of this pathology. Nevertheless, lack of consensus exists in the pursuit of a predictable therapy. Different therapeutic modalities have been advocated. Non-surgical therapy as a sole modality is often insufficient to resolve inflammation. Surgical interventions have demonstrated more favorable outcomes. Amongst these, evidence supported the application of resective, reconstructive, or combined approaches to limit progressive bone loss and achieve soft tissue health. Nevertheless, up to date, the most suitable modality remains unknown and the decision-making process derives from the understanding acquired from the management of periodontitis.

One critical element regarded to successfully resolve peri-implantitis is to efficiently detoxify the contaminated implant surface. Mechanical, pharmacological and chemical strategies have been proposed to eliminate bacterial plaque and remnants from the implant surface. However, evidence has not demonstrated superiority of a given detoxification agent/strategy.

In this sense, the significance of barrier membranes is not yet well understood. Roos-Jansaker in 2014 showed that the additional use of barrier membranes did not improve the outcome. Nevertheless, since then this subject has not been a matter of research.

DETAILED DESCRIPTION:
The effect of barrier membrane in the reconstructive management of peri-implantitis will be tested at 12-month follow-up

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers
* No use of antibiotics recently
* No metabolic disorder
* Infra-osseous or combined peri-implantitis defect

Exclusion Criteria:

* Smokers
* Pregnant
* Metabolic disorders that affect bone healing
* Supra-crestal defects

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
Changes in clinical parameters | 12 months
  Number of patients where the disease was resolved. At implant level the changes in bleeding on probing and changes in probing pocket depths will be recorded as well

SECONDARY OUTCOMES:
Changes in Bone level | 12-month follow-up
  Change in Bone level measured in mm from x-rays obtained from the comparative between baseline bone level and bone level determined at 12-month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica CICOM, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: Undecided
To publish once collected the data

REFERENCES:
- [Background] Monje A, Pons R, Roccuzzo A, Salvi GE, Nart J. Reconstructive therapy for the management of peri-implantitis via submerged guided bone regeneration: A prospective case series. Clin Implant Dent Relat Res. 2020 Jun;22(3):342-350. doi: 10.1111/cid.12913. Epub 2020 May 14. PMID 32410379
- [Result] Monje A, Pons R, Amerio E, Wang HL, Nart J. Resolution of peri-implantitis by means of implantoplasty as adjunct to surgical therapy: A retrospective study. J Periodontol. 2022 Jan;93(1):110-122. doi: 10.1002/JPER.21-0103. Epub 2021 May 15. PMID 33904175
- [Derived] Monje A, Pons R, Vilarrasa J, Nart J, Wang HL. Significance of barrier membrane on the reconstructive therapy of peri-implantitis: A randomized controlled trial. J Periodontol. 2023 Mar;94(3):323-335. doi: 10.1002/JPER.22-0511. Epub 2022 Dec 12. PMID 36399349